CLINICAL TRIAL: NCT04595708
Title: Telephone Calls for Health for Homebound Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Collaborators: Meals on Wheels Central Texas (Other)
Responsible Party: Principal Investigator, Maninder Kahlon, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-05-0009
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Loneliness; Social Isolation; Depression
MeSH Terms: conditions — Social Isolation; Depression

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The individual who collected baseline and follow-up surveys was blinded to the status of the participant as part of control or intervention group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention - Calls (Experimental): Participants randomized to the intervention will receive a call of between 5 - 10 minutes in length each by a consistent caller, five times a week, Monday through Friday for 4 consecutive weeks to check in on them. After the first week of calls, subjects in the intervention arm will be asked if the frequency of calls is acceptable or if they would like to reduce the call frequency, potentially to a minimum of twice per week.
  Interventions: Behavioral: Phone Call
- Control - No calls (No Intervention): Participants randomized to a control group will not receive the intervention calls. The control group will receive calls from a member of the research team at the beginning of the study to collect baseline survey data and at the post-4-week period to collect post-study survey data.

INTERVENTIONS:
Behavioral: Phone Call — Calls were made by volunteers trained to engage with participants. Call structure was unscripted and call length was recommended to be between 5-10 min.
  Arms: Intervention - Calls

SUMMARY:
A randomized controlled trial of the effect of 4 weeks of regular check-in calls, up to 5 per week based on participant's choice and 2 survey collection calls and possible referral of other services, versus no daily check-in calls, on self-reported loneliness measures for current Meals on Wheels participants (MOW).

DETAILED DESCRIPTION:
The intervention arm will include 125 MOW clients to receive a call of between 5 - 10 minutes in length each by a consistent caller, five times a week, Monday through Friday for 4 consecutive weeks to check in on them. After the first week of calls, subjects in the intervention arm will be asked if the frequency of calls is acceptable or if they would like to reduce the call frequency, potentially to a minimum of twice per week.

Brief guidance and training will be provided for the daily conversation to maximize time spent speaking by the recipient but otherwise, the calls are unscripted other than specific prompts to ask about the recipient's general sense of well-being. "How are you doing today?"

The control Arm will include 125 MOW clients who will be randomized to a control group that will not receive the intervention calls. The control group will receive calls from a member of the research team at the beginning of the study to collect baseline survey data and at the post-4-week period to collect post-study survey data.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18+) clients of Meals on Wheels of Central Texas

Exclusion Criteria:

* Cognitive impairment or in a hospice program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-26 (Actual)

PRIMARY OUTCOMES:
Loneliness as assessed by the De Jong Gierveld Loneliness Scale | 4 weeks
  Investigators will use the De Jong Gierveld Loneliness 6-Item Scale for Overall, Emotional, and Social Loneliness. Scored from 0-6, a score of 0 indicates least lonely while a score of 6 indicates most lonely.
Loneliness as Assessed by the UCLA Short Scale for Measuring Loneliness in Large Surveys | 4 weeks
  Investigators will use the UCLA Short Scale for Measuring Loneliness in Large Surveys to measure loneliness. Scored from 3-9, higher scores indicate greater degrees of loneliness.

SECONDARY OUTCOMES:
Depression as Assessed by the 8-item Depression Health Questionnaire (PHQ-8) | 4 weeks
  Investigators will use the Depression Patient Health Questionnaire (PHQ-8) to measure depression. Scored from 0-3, and a score of 0 indicates lower levels of depression while a score of 3 indicates higher levels of depression.
Anxiety as Assessed by the 7-item Generalized Anxiety Disorder Scale (GAD-7) | 4 weeks
  Investigators will use the Generalized Anxiety Disorder Scale (GAD-7) to measure anxiety. Scored from 0-3, and a score of 0 indicates lower levels of anxiety while a score of 3 indicates higher levels of anxiety.
Health Status and Quality of Life as Assessed by the Short Form-12 Question Survey | 4 weeks
  Investigators will use the Short Form-12 question survey to measure physical and mental health status. Summary scores range from 0-100, with higher scores indicating a better self-reported level of health.
Social Engagement as Assess by the Short Lubben Social Network Scale (LSNS) | 4 weeks
  Investigators will use the 6-item Short Lubben Social Network Scale to measure social engagement. For the LSNS-6, the score ranges between 0 and 30, with a higher score indicating more social engagement.
Empathy as Assessed by The Consultation and Relational Empathy (CARE) Measure | After the 4 week intervention (follow-up)
  Investigators will use the CARE Measure to evaluate measures of empathy in the context of the caller/participant relationship
Toronto Empathy Questionnaire | Prior to the 4 week intervention (baseline)
  The Toronto Empathy Questionnaire will be used to assess characteristics of callers that align with measures of ability to be empathetic.

CONTACTS AND LOCATIONS:
Overall Officials: Maninder Kahlon, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holt-Lunstad J, Smith TB, Baker M, Harris T, Stephenson D. Loneliness and social isolation as risk factors for mortality: a meta-analytic review. Perspect Psychol Sci. 2015 Mar;10(2):227-37. doi: 10.1177/1745691614568352. PMID 25910392
- [Background] Anderson, G., Thayer, C. . Loneliness and Social Connections: A National Survey of Adults 45 and Older. Washington, DC: AARP Research, September 2018. https://doi.org/10.26419/res.00246.001.
- [Background] Cacioppo JT, Hughes ME, Waite LJ, Hawkley LC, Thisted RA. Loneliness as a specific risk factor for depressive symptoms: cross-sectional and longitudinal analyses. Psychol Aging. 2006 Mar;21(1):140-51. doi: 10.1037/0882-7974.21.1.140. PMID 16594799
- [Background] Steger MF, Kashdan TB. Depression and Everyday Social Activity, Belonging, and Well-Being. J Couns Psychol. 2009 Apr;56(2):289-300. doi: 10.1037/a0015416. PMID 20428460
- [Background] Derksen F, Bensing J, Lagro-Janssen A. Effectiveness of empathy in general practice: a systematic review. Br J Gen Pract. 2013 Jan;63(606):e76-84. doi: 10.3399/bjgp13X660814. PMID 23336477
- [Derived] Kahlon MK, Aksan N, Aubrey R. Effect of a Layperson-Delivered Telephone Program for People With Depressive Symptoms. Psychiatr Serv. 2023 Nov 1;74(11):1176-1179. doi: 10.1176/appi.ps.20220440. Epub 2023 Apr 12. PMID 37042110
- [Derived] Kahlon MK, Aksan N, Aubrey R, Clark N, Cowley-Morillo M, Jacobs EA, Mundhenk R, Sebastian KR, Tomlinson S. Effect of Layperson-Delivered, Empathy-Focused Program of Telephone Calls on Loneliness, Depression, and Anxiety Among Adults During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Psychiatry. 2021 Jun 1;78(6):616-622. doi: 10.1001/jamapsychiatry.2021.0113. PMID 33620417